CLINICAL TRIAL: NCT04870866
Title: NAD Supplementation to Prevent Progressive Neurological Disease in Ataxia Telangiectasia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: The Bergesen Foundation (Other); South-Eastern Norway Regional Health Authority (Other); Sykehuset Innlandet HF (Other); Oslo University Hospital (Other); St. Olavs Hospital (Other); Haukeland University Hospital (Other); University Hospital of North Norway (Other); University of Bergen (Other)
Responsible Party: Principal Investigator, Hilde Nilsen, Professor, University Hospital, Akershus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/419
Record Dates: First submitted 2021-04-23; First posted 2021-05-04 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Ataxia Telangiectasia
Keywords: ataxia telangiectasia; nicotinamide ribonucleoside; Louis-Bar syndrome
MeSH Terms: conditions — Ataxia Telangiectasia | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Open label proof of concept
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- NR treated (Experimental): Nicotinamide ribonuceloside (NR), sold under the trade name Niagen™
  Interventions: Drug: Nicotinamide ribonucleoside

INTERVENTIONS:
Drug: Nicotinamide ribonucleoside — Two year intervention
  Other Names: Niagen

SUMMARY:
The study investigates the effect of dietary supplementation of nicotinamide ribonucleoside (NR) in children with ataxia telangiectasia (AT), with main focus on neurological symptoms.

DETAILED DESCRIPTION:
Ataxia Telangiectasia (AT) is a genetic disease, where patients are born with mutations in the Ataxia- Telangiectasia Mutated (ATM) gene. The gene codes for the ATM kinase, which is required for repair of DNA double-stranded breaks and DNA damage response signalling.

There is no treatment available for the neurological manifestations of AT.

The study investigates the effects of NR (300 mg/day) during 2 years.

ELIGIBILITY:
Inclusion Criteria:

* clinically and molecular verified classical A-T disease

Exclusion Criteria:

* less than 2 years of age
* participation in other on-going study
* pregnancy
* liver failure
* other severe medical conditions considered to set patient at risk

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2024-09-03 (Estimated); Study Completion 2027-06-16 (Estimated)

PRIMARY OUTCOMES:
NAD metabolome | 2 years
  Increase of NAD+ and other stable NAD+ metabolites (referred to as the NAD metabolome) in blood

SECONDARY OUTCOMES:
Patient well being | 2 years
  Improved or stabilized health-related quality of life (HRQOL) measured with the Pediatric Quality of Life Inventory (PedSQL)
Motoric function - The Scale for the Assessment and Rating of Ataxia (SARA) | 2 years
  Stabilized motoric function measured with SARA.
  The SARA scale is made up of measurements related to gait, stance, sitting, speech, finger-chase test, nose-finger test, fast alternating movements and heel-shin test.
  The range is from no ataxia (value 0) to severe ataxia (value 40).
Motoric function - The International Cooperative Ataxia Rating Scale (ICARS) | 2 years
  Stabilized motoric function measured with ICARS.
  The ICARS scale is made from measurements of postural and gait disturbances, limb ataxia, dysarthria, and oculomotor disorders.
  The range is from no ataxia (value 0) to severe ataxia (value 100).
Motoric function - Customized gait scale (GS) | 2 years
  Stabilized motoric function measured with GS.
  The gait scale assess gait functionality in patients with Ataxia-telangiectasia.
  The range is from no walking ability (value 0) to normal walking ability according to age and maturity (value 10).
Motoric function - AT Neuro Examination Scale Toolkit, updated version (AT-NEST) | 2 years
  Stabilized motoric function measured with AT-NEST.
  The AT-NEST scale is made from scoring of speech, handwriting/drawing, oculomotor, ataxia, muscle strength, neuropathy, growth, nutrition, learning ability/cognition, MS mental state.
  The range is from normal (value 144) to severe ataxia (value 0).
Motoric function - Clinical Global Scale rating instrument for A-T | 2 years
  Stabilized motoric function measured with Clinical Global Scale rating instrument for A-T.
  The Clinical Global Scale rating instrument for A-T scale is made from scoring of gait ataxia, dysmetria, dysarthria, extrapyramidal movements and eye movements.
  The range is from normal (value 0) to severe (value 4).
Liver function | 2 years
  Normalized or stabilized liver function as assessed by blood levels of
  -alfa fetoprotein (AFP)
Blood sugar control | 2 years
  Normalized or stabilized blood sugar levels as measured in blood:
  -HbA1c
Mitochondrial function | 2 years
  Normalized or stabilized mitochondrial markers in blood:
  * lactate
  * lactate dehydrogenase
  * FGF21

CONTACTS AND LOCATIONS:
Overall Officials: Hilde L Nilsen, Principal Investigator — University Hospital, Akershus
Locations (2):
- Norway (2):
  - Hilde Loge Nilsen, Lørenskog
  - Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fang EF, Kassahun H, Croteau DL, Scheibye-Knudsen M, Marosi K, Lu H, Shamanna RA, Kalyanasundaram S, Bollineni RC, Wilson MA, Iser WB, Wollman BN, Morevati M, Li J, Kerr JS, Lu Q, Waltz TB, Tian J, Sinclair DA, Mattson MP, Nilsen H, Bohr VA. NAD+ Replenishment Improves Lifespan and Healthspan in Ataxia Telangiectasia Models via Mitophagy and DNA Repair. Cell Metab. 2016 Oct 11;24(4):566-581. doi: 10.1016/j.cmet.2016.09.004. PMID 27732836